CLINICAL TRIAL: NCT01353911
Title: A Randomized, Active-Controlled, Dose-Ranging Estimation Study to Evaluate the Safety, Tolerability, and Efficacy of Different Regimens of MK-5172 When Administered Concomitantly With Peginterferon Alfa-2b and Ribavirin in Treatment-Naïve Patients With Chronic Genotype 1 Hepatitis C Virus Infection
Brief Title: Grazoprevir (MK-5172) Administered With Peginterferon and Ribavirin in Treatment-Naïve Participants With Chronic Hepatitis C (MK-5172-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-003; 2011-000759-18 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Grazoprevir 100 mg (Experimental): TN non-cirrhotic (NC) participants receive Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Grazoprevir; Drug: Placebo for Boceprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Grazoprevir 200 mg (Experimental): TN NC participants receive Grazoprevir 200 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Grazoprevir; Drug: Placebo for Boceprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Grazoprevir 400 mg (Experimental): TN NC participants receive Grazoprevir 400 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Grazoprevir; Drug: Placebo for Boceprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Grazoprevir 800 mg (Experimental): TN NC participants receive Grazoprevir 800 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Grazoprevir; Drug: Placebo for Boceprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Boceprevir 800 mg (Active Comparator): TN NC participants start a 4 week lead-in with Peg-IFN + RBV, then receive Boceprevir 800 mg + Peg-IFN + RBV for 24 weeks followed by 0 or 20 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Boceprevir; Drug: Placebo for Grazoprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Grazoprevir 400 mg/100 mg (Experimental): As the result of an interim analysis, TN NC participants assigned to the 400 mg grazoprevir group were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV and will remain in the study.
  Interventions: Drug: Grazoprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- Grazoprevir 800 mg/100 mg (Experimental): As the result of an interim analysis, TN NC participants assigned to the 800 mg grazoprevir group were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV and will remain in the study.
  Interventions: Drug: Grazoprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin
- OL Grazoprevir 100 mg (Experimental): TN cirrhotic participants receive open-label Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
  Interventions: Drug: Grazoprevir; Drug: Peg-interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Grazoprevir — Orally once daily in AM. Blinded or open-label depending on treatment arm.
  Arms: Grazoprevir 100 mg; Grazoprevir 200 mg; Grazoprevir 400 mg; Grazoprevir 400 mg/100 mg; Grazoprevir 800 mg; Grazoprevir 800 mg/100 mg; OL Grazoprevir 100 mg
Drug: Boceprevir — Four 200 mg capsules orally three times daily.
  Other Names: Victrelis
  Arms: Boceprevir 800 mg
Drug: Placebo for Grazoprevir — Orally once daily in AM.
  Arms: Boceprevir 800 mg
Drug: Placebo for Boceprevir — Four capsules orally three times daily.
  Arms: Grazoprevir 100 mg; Grazoprevir 200 mg; Grazoprevir 400 mg; Grazoprevir 800 mg
Drug: Peg-interferon alfa-2b — 1.5 μg/kg/week subcutaneous injection.
  Other Names: PegIntron; Peg-IFN alfa-2b
Drug: Ribavirin — 300 mg to 700 mg orally twice daily.
  Other Names: Rebetol

SUMMARY:
This study will evaluate the safety, tolerability, and antiviral activity of grazoprevir (MK-5172) when administered in combination with peginterferon alfa-2b (Peg-IFN) and ribavirin (RBV) in treatment-naïve (TN) participants with chronic hepatitis C.

DETAILED DESCRIPTION:
Amendment 4 unblinded treatment after an interim analysis for all subsequently enrolled TN participants (the Second Cohort) who were receiving grazoprevir 400 or 800 mg daily, and they were down-dosed to 100 mg daily between Treatment Week (TW) 3 and TW12 for the remainder of the 12-week treatment course.

Amendment 5 allowed treatment-naïve participants with chronic hepatitis C and compensated cirrhosis to be enrolled and receive open-label grazoprevir 100 mg in combination with Peg-IFN and RBV, without a corresponding control arm.

ELIGIBILITY:
Inclusion Criteria:

* Has previously documented chronic hepatitis C genotype 1 (CHC GT 1) infection
* Has hepatitis C virus (HCV) ribonucleic acid (RNA value) ≥10,000 IU/mL
* Body weight ≥40 kg (88 lbs) and ≤125 kg (275 lbs)
* Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs and symptoms of decompensated liver disease
* Had a liver biopsy within 3 years of screening or between screening and Day 1 with histology consistent with CHC and no evidence of cirrhosis or hepatocellular carcinoma or no other cause for chronic liver disease (for participants with compensated cirrhosis, any liver biopsy demonstrating cirrhosis regardless of length of time since biopsy)
* Female of childbearing potential or a male with female sexual partner who is of childbearing potential agrees to use two acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations
* For participants with compensated cirrhosis, evidence of cirrhosis without evidence of hepatocellular carcinoma (confirmed by ultrasound within 4 weeks prior)

Exclusion Criteria:

* Is pregnant, breastfeeding, or plans to become pregnant or donate eggs
* Is human immunodeficiency virus (HIV) positive or known to be co-infected with hepatitis B virus
* Has received prior approved or investigational treatment for hepatitis C
* Has evidence of hepatocellular carcinoma or is under evaluation for hepatocellular carcinoma
* For participants with compensated cirrhosis: alphafetoprotein level of ≥100 ng/mL
* Has evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years
* Has evidence or history of chronic hepatitis not caused by HCV
* Is diabetic and/or hypertensive with clinically significant ocular examination findings: retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or any other clinically significant abnormality
* Has any known medical condition that could interfere with participation in and completion of the study
* Pre-existing psychiatric condition including but not limited to moderate or severe depression, suicidal or homicidal ideation or attempt, schizophrenia, psychosis, bipolar disorder, post traumatic stress disorder, or mania
* Is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent
* Member or family member of study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2013-01-20 (Actual); Study Completion 2015-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Manns MP, Vierling JM, Bacon BR, Bruno S, Shibolet O, Baruch Y, Marcellin P, Caro L, Howe AY, Fandozzi C, Gress J, Gilbert CL, Shaw PM, Cooreman MP, Robertson MN, Hwang P, Dutko FJ, Wahl J, Mobashery N. The combination of MK-5172, peginterferon, and ribavirin is effective in treatment-naive patients with hepatitis C virus genotype 1 infection without cirrhosis. Gastroenterology. 2014 Aug;147(2):366-76.e6. doi: 10.1053/j.gastro.2014.04.006. Epub 2014 Apr 12. PMID 24727022
- [Derived] Howe AY, Black S, Curry S, Ludmerer SW, Liu R, Barnard RJ, Newhard W, Hwang PM, Nickle D, Gilbert C, Caro L, DiNubile MJ, Mobashery N. Virologic resistance analysis from a phase 2 study of MK-5172 combined with pegylated interferon/ribavirin in treatment-naive patients with hepatitis C virus genotype 1 infection. Clin Infect Dis. 2014 Dec 15;59(12):1657-65. doi: 10.1093/cid/ciu696. Epub 2014 Sep 28. PMID 25266289

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 368 participants enrolled on study. 36 cirrhotic participants received open-label (OL) grazoprevir + peginterferon (Peg-IFN) + ribavirin (RBV), and 332 non-cirrhotic participants were randomized to receive 100, 200, 400, or 800 mg grazoprevir + Peg-IFN + RBV. 43 in the 400 mg group and 36 in the 800 mg group were down-dosed to 100 mg grazoprevir.
Groups:
- OL Grazoprevir 100 mg: Treatment-naïve (TN) cirrhotic participants received open-label Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 100 mg: TN non-cirrhotic (NC) participants received Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 200 mg: TN NC participants received Grazoprevir 200 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 400 mg: TN NC participants received Grazoprevir 400 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 800 mg: TN NC participants received Grazoprevir 800 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 400 mg/100 mg: TN NC participants initially were randomized to receive Grazoprevir 400 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy. As the result of an interim analysis, these participants were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Grazoprevir 800 mg/100 mg: TN NC participants initially were randomized to receive Grazoprevir 800 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy. As the result of an interim analysis, these participants were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Boceprevir 800 mg: TN NC participants started a 4 week lead-in with Peg-IFN + RBV, then received Boceprevir 800 mg + Peg-IFN + RBV for 24 weeks followed by 0 or 20 weeks of Peg-IFN + RBV, based on response guided therapy.
Period: Overall Study
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Started | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
Completed | 28 | 57 | 59 | 22 | 23 | 36 | 30 | 51
Not Completed | 8 | 9 | 9 | 2 | 6 | 7 | 6 | 15
Not completed — Lost to Follow-up | 2 | 6 | 4 | 0 | 4 | 4 | 3 | 6
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 2 | 2 | 3 | 3 | 9
Not completed — Status Not Recorded | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS); all randomized/enrolled participants who received ≥1 dose of study treatment. Results for participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens.
Groups:
- Grazoprevir 100 mg: TN NC participants received Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Total: Total of all reporting groups
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg | Total
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (6.9) | 46.4 (11.3) | 48.3 (10.6) | 44.6 (12.5) | 50.4 (13.4) | 48.3 (11.4) | 50.3 (11.2) | 48.3 (11.2) | 48.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 25 | 32 | 12 | 15 | 15 | 13 | 29 | 155
  Male | 22 | 41 | 36 | 12 | 14 | 28 | 23 | 37 | 213

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Early Viral Response (cEVR)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). cEVR was defined as undetectable HCV RNA (target not detected [TND]) at Week 12. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: After 12 weeks of treatment with grazoprevir/boceprevir
Population: FAS; all randomized/enrolled participants who received ≥1 dose of study treatment. A Missing = Failure approach was used for missing data. Results for participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
percentage of participants | 94.4 [81.3 to 99.9] | 80.3 [68.7 to 89.1] | 85.3 [74.6 to 92.7] | 87.5 [67.6 to 97.3] | 75.9 [56.5 to 89.7] | 86.0 [72.1 to 94.7] | 86.1 [70.5 to 95.3] | 69.7 [57.1 to 80.4]

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) During the Treatment Period and First 14 Follow-up Days
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE.
Time Frame: Treatment period plus the first 14 days of follow-up (up to 50 weeks)
Population: All Participants as Treated (APaT) population; all randomized/enrolled who received ≥1 dose of study treatment according to treatment actually received. Participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens.
Measure: Number; unit: participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
participants | 34 | 65 | 66 | 23 | 28 | 42 | 35 | 64

3. Primary Outcome: Number of Participants Who Discontinued Study Medication Due to AEs During the Treatment Period and First 14 Follow-up Days
Description: as for outcome 2
Time Frame: Treatment period plus the first 14 days of follow-up (up to 50 weeks)
Population: APaT population; all randomized/enrolled who received ≥1 dose of study treatment according to treatment actually received. Participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens.
Measure: Number; unit: participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
participants | 2 | 3 | 4 | 2 | 3 | 4 | 2 | 9

4. Secondary Outcome: Median Time to First Achievement of Undetectable HCV RNA During Treatment
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. Undetectable HCV RNA (target not detected [TND]) was defined as below the 9.3 IU/ml limit of detection. Kaplan Meier summary statistics were calculated for each treatment arm.
Time Frame: From first dose of study medication until first achievement of undetectable HCV RNA (up to 48 weeks of treatment)
Population: FAS; all randomized/enrolled participants who received ≥1 dose of study treatment. Results for participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens. Participants in the FAS not achieving TND were censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
days | 22.0 [21.0 to 29.0] | 15.0 [15.0 to 18.0] | 28.0 [23.0 to 29.0] | 16.0 [14.0 to 29.0] | 16.5 [14.0 to 28.0] | 27.0 [15.0 to 29.0] | 29.0 [15.0 to 29.0] | 57.0 [57.0 to 59.0]

5. Secondary Outcome: Percentage of Participants Achieving Rapid Viral Response (RVR)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). RVR was defined as undetectable (TND) HCV RNA at Week 4 of study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: After 4 weeks of treatment with grazoprevir/boceprevir
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
percentage of participants | 72.2 [54.8 to 85.8] | 90.9 [81.3 to 96.6] | 91.2 [81.8 to 96.7] | 87.5 [67.6 to 97.3] | 86.2 [68.3 to 96.1] | 81.4 [66.6 to 91.6] | 83.3 [67.2 to 93.6] | 59.1 [46.3 to 71.0]

6. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of Study Therapy (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). SVR12 was defined as undetectable (TND) HCV RNA at 12 weeks after the end of all study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: 12 weeks after the end of all treatment (up to 60 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
percentage of participants | 72.2 [54.8 to 85.8] | 89.4 [79.4 to 95.6] | 91.2 [81.8 to 96.7] | 87.5 [67.6 to 97.3] | 79.3 [60.3 to 92.0] | 93.0 [80.9 to 98.5] | 91.7 [77.5 to 98.2] | 60.6 [47.8 to 72.4]

7. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of Study Therapy (SVR24)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). SVR24 was defined as undetectable (TND) HCV RNA at 24 weeks after the end of all study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: 24 weeks after the end of all treatment (up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
percentage of participants | 72.2 [54.8 to 85.8] | 86.4 [75.7 to 93.6] | 92.6 [83.7 to 97.6] | 87.5 [67.6 to 97.3] | 79.3 [60.3 to 92.0] | 93.0 [80.9 to 98.5] | 91.7 [77.5 to 98.2] | 57.6 [44.8 to 69.7]

8. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA at Week 72
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. Undetectable HCV RNA (target not detected [TND]) was defined as below the 9.3 IU/ml limit of detection. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Grazoprevir 100 mg | Grazoprevir 100 mg | Grazoprevir 200 mg | Grazoprevir 400 mg | Grazoprevir 800 mg | Grazoprevir 400 mg/100 mg | Grazoprevir 800 mg/100 mg | Boceprevir 800 mg
Number analyzed (Participants) | 36 | 66 | 68 | 24 | 29 | 43 | 36 | 66
percentage of participants | 69.4 [51.9 to 83.7] | 80.3 [68.7 to 89.1] | 86.8 [76.4 to 93.8] | 87.5 [67.6 to 97.3] | 75.9 [56.5 to 89.7] | 79.1 [64.0 to 90.0] | 83.3 [67.2 to 93.6] | 54.5 [41.8 to 66.9]

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to 72 weeks
Description: APaT population; all randomized/enrolled who received ≥1 dose of study treatment according to treatment actually received. Participants who received grazoprevir 400 or 800 mg and were then down-dosed to receive grazoprevir 100 mg are reported separately from participants who completed the 400 mg and 800 mg regimens.
Groups:
- Cirr: OL Grazoprevir 100 mg: TN cirrhotic participants received open-label Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 100 mg: TN NC participants received Grazoprevir 100 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 200 mg: TN NC participants received Grazoprevir 200 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 400 mg: TN NC participants received Grazoprevir 400 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 800 mg: TN NC participants received Grazoprevir 800 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 400 mg/100 mg: TN NC participants initially were randomized to receive Grazoprevir 400 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy. As the result of an interim analysis, these participants were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Grazoprevir 800 mg/100 mg: TN NC participants initially were randomized to receive Grazoprevir 800 mg + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy. As the result of an interim analysis, these participants were unblinded and transitioned to 100 mg grazoprevir once daily + Peg-IFN + RBV for 12 weeks followed by 12 or 36 weeks of Peg-IFN + RBV, based on response guided therapy.
- Non-cirr: Boceprevir 800 mg: TN NC participants started a 4 week lead-in with Peg-IFN + RBV, then received Boceprevir 800 mg + Peg-IFN + RBV for 24 weeks followed by 0 or 20 weeks of Peg-IFN + RBV, based on response guided therapy.
Arm/Group | Cirr: OL Grazoprevir 100 mg | Non-cirr: Grazoprevir 100 mg | Non-cirr: Grazoprevir 200 mg | Non-cirr: Grazoprevir 400 mg | Non-cirr: Grazoprevir 800 mg | Non-cirr: Grazoprevir 400 mg/100 mg | Non-cirr: Grazoprevir 800 mg/100 mg | Non-cirr: Boceprevir 800 mg
Serious Adverse Events (participants affected / at risk) | 3/36 | 6/66 | 9/68 | 2/24 | 2/29 | 5/43 | 4/36 | 5/66
Other Adverse Events (participants affected / at risk) | 34/36 | 64/66 | 65/68 | 23/24 | 27/29 | 42/43 | 36/36 | 64/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirr: OL Grazoprevir 100 mg (N=36) | Non-cirr: Grazoprevir 100 mg (N=66) | Non-cirr: Grazoprevir 200 mg (N=68) | Non-cirr: Grazoprevir 400 mg (N=24) | Non-cirr: Grazoprevir 800 mg (N=29) | Non-cirr: Grazoprevir 400 mg/100 mg (N=43) | Non-cirr: Grazoprevir 800 mg/100 mg (N=36) | Non-cirr: Boceprevir 800 mg (N=66)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Segmented hyalinising vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirr: OL Grazoprevir 100 mg (N=36) | Non-cirr: Grazoprevir 100 mg (N=66) | Non-cirr: Grazoprevir 200 mg (N=68) | Non-cirr: Grazoprevir 400 mg (N=24) | Non-cirr: Grazoprevir 800 mg (N=29) | Non-cirr: Grazoprevir 400 mg/100 mg (N=43) | Non-cirr: Grazoprevir 800 mg/100 mg (N=36) | Non-cirr: Boceprevir 800 mg (N=66)
Anaemia (Blood and lymphatic system disorders) | 13 (16) | 11 (16) | 17 (21) | 2 (2) | 7 (7) | 5 (7) | 7 (7) | 18 (25)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 5 (9)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 6 (12) | 7 (8) | 2 (3) | 1 (2) | 2 (3) | 0 (0) | 11 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3) | 7 (8) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 7 (7) | 5 (6) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 11 (13) | 11 (13) | 5 (6) | 11 (14) | 5 (5) | 12 (13) | 16 (19)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 7 (7) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 9 (10) | 25 (29) | 25 (28) | 6 (8) | 16 (21) | 15 (17) | 19 (29) | 31 (37)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Toothache (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 8 (13) | 8 (10) | 6 (8) | 5 (7) | 4 (9) | 6 (7) | 16 (20)
Asthenia (General disorders) | 8 (9) | 14 (19) | 9 (9) | 5 (5) | 3 (4) | 7 (8) | 8 (8) | 12 (13)
Chest pain (General disorders) | 4 (4) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Chills (General disorders) | 10 (11) | 20 (22) | 19 (20) | 6 (7) | 10 (10) | 12 (12) | 11 (12) | 15 (16)
Fatigue (General disorders) | 18 (19) | 27 (30) | 31 (38) | 11 (12) | 16 (19) | 17 (17) | 15 (16) | 27 (30)
Influenza like illness (General disorders) | 9 (9) | 14 (15) | 20 (22) | 7 (7) | 5 (5) | 15 (15) | 7 (7) | 23 (24)
Injection site erythema (General disorders) | 2 (2) | 12 (12) | 10 (10) | 1 (1) | 8 (8) | 2 (2) | 3 (3) | 8 (9)
Injection site irritation (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Injection site reaction (General disorders) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 8 (8) | 12 (13) | 12 (12) | 3 (3) | 11 (11) | 8 (8) | 4 (4) | 12 (13)
Pyrexia (General disorders) | 9 (9) | 20 (23) | 24 (27) | 12 (12) | 8 (10) | 12 (18) | 6 (22) | 20 (21)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 4 (6) | 8 (8) | 3 (3) | 6 (6) | 3 (5) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (8)
Spleen palpable (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 5 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 16 (17) | 11 (11) | 4 (5) | 9 (9) | 10 (10) | 14 (14) | 15 (16)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (11) | 9 (13) | 7 (8) | 4 (7) | 3 (3) | 7 (7) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 4 (4) | 0 (0) | 2 (3) | 2 (2) | 5 (7) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 12 (13) | 9 (11) | 6 (9) | 4 (5) | 7 (7) | 5 (6) | 13 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 4 (4) | 8 (9) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8) | 6 (6) | 10 (10) | 2 (2) | 6 (6) | 5 (6) | 5 (6) | 9 (9)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5) | 7 (7) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 19 (19)
Headache (Nervous system disorders) | 12 (16) | 28 (39) | 31 (35) | 8 (8) | 12 (16) | 12 (13) | 17 (19) | 35 (44)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (4)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Poor quality sleep (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 5 (5) | 10 (10) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 7 (7) | 11 (11) | 1 (1) | 5 (5) | 6 (6) | 8 (8) | 7 (7)
Insomnia (Psychiatric disorders) | 8 (10) | 15 (15) | 10 (10) | 3 (3) | 6 (7) | 7 (7) | 8 (10) | 21 (22)
Irritability (Psychiatric disorders) | 10 (10) | 16 (16) | 9 (11) | 1 (1) | 3 (3) | 7 (7) | 5 (7) | 12 (14)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 9 (9) | 1 (1) | 4 (5) | 9 (10) | 6 (6) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (8) | 10 (12) | 1 (1) | 3 (5) | 2 (2) | 4 (4) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 6 (7) | 0 (0) | 6 (6) | 6 (6) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 6 (7) | 2 (2) | 4 (4) | 1 (1) | 3 (3) | 6 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 17 (17) | 19 (20) | 7 (7) | 9 (10) | 8 (8) | 10 (10) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 9 (10) | 1 (1) | 2 (2) | 7 (7) | 5 (5) | 8 (8)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 12 (16) | 15 (17) | 6 (6) | 7 (7) | 4 (4) | 10 (11) | 10 (12)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 15 (17) | 13 (14) | 3 (7) | 6 (7) | 7 (12) | 9 (10) | 17 (22)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (4) | 2 (7) | 1 (3) | 1 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.